Ouality of Recovery after Dexamethasone, Ondansetron or Placebo Intrathecal

Morphine Administration

NCT03035942

February 1st, 2018

Statistical analysis

The primary outcome was the QoR-40 score 24 hours after surgery. Murphy et al

evaluated the quality of recovery in patients undergoing laparoscopic cholecystectomy

with or without IV dexamethasone. The sample size estimated to achieve 80% power

to detect a 17-point difference in QoR-40 was 30 subjects per group. A difference of 10

points represents a 15% improvement in the quality of recovery. <sup>2,3</sup>Considering possible

dropouts, one hundred thirty-five subjects were finally randomized into three groups.

The Shapiro-Wilk test was used to test the hypothesis of a normal distribution. Ordinal

and continuous data that were not normally distributed are presented as median and

range and were compared using the Kruskal-Wallis test. Dunn's multiple comparisons

test was used to compare groups whenever a difference was detected. Treatment

comparisons were tested at a 1.67% level (Bonferroni comparison). Statistical

significance (p-value) was assessed by means of a two-tailed test in all instances; values

below 0.05 were considered statistically significant. Statistical analysis was performed

using O IBM SPSS Statistics, version 22.

1. Murphy GS, Szokol JW, Greenberg SB, Avram MJ, Vender JS, Nisman M,

Vaughn J. Preoperative dexamethasone enhances quality of recovery after

- laparoscopic cholecystectomy: effect on in-hospital and postdischarge recovery outcomes. Anesthesiology 2011; 114: 882-90.
- 2. Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Vality and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000; 84:11-15.
- 3. Castro-Alves LJS, de Azevedo VFL, Braga TFF, Gonçalves AC, de Oliveira GS. The effect of neuroaxial versus general anesthesia techniques on postoperative quality and analgesia after abdominal hysterectomy: a prospective, randomized, controlled trial. Anesth Analg 2011; 113: 1480-6